CLINICAL TRIAL: NCT06679062
Title: A Double-masked, Randomized, Phase II Study to Compare the Effectiveness of 20mg Oral Suvorexant (SUV) Versus Placebo (1:1) in Participants With Co-occurring Alcohol Use Disorder (AUD) and Posttraumatic Stress Disorder (PTSD)
Brief Title: Suvorexant for Treatment of AUD and PTSD
Acronym: SUV
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacotherapies for Alcohol and Substance Use Disorders Alliance (Other)
Collaborators: University of California, Los Angeles (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AS210006-A10
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Use Disorder (AUD); Post Traumatic Stress Disorder (PTSD); Insomnia
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders | interventions — suvorexant; Orexin Receptor Antagonists

STUDY DESIGN:
Intervention Model Description: Each participant will be given a placebo run-in (Day -7 to Day -1). On baseline (Day 0), the participant will be randomized to receive SUV or placebo (1:1 ratio) and administered 10mg SUV or placebo for an additional 7 days (Day 0 to Day 6). On Day 7, the participant previously randomized to SUV will be given 20 mg SUV, and participant previously randomized to placebo will continue with placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: To minimize bias, all participants will be screened for assurance that they meet study eligibility criteria. A placebo drug will be employed as the comparison group to active study drug and the study will be conducted in a double-blinded fashion in that both the participants and the site investigators and staff interacting with participants and assessing study outcomes will be blinded to treatment assignment. The only individuals at the site with access to treatment assignment information will be the research pharmacists.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 10mg and 20mg Suvorexant (SUV) (Active Comparator): Participants will be randomly assigned to receive SUV (10mg (Days 0-6) and 20mg (Days 7-13)).
  Interventions: Drug: Suvorexant
- Placebo (Placebo Comparator): Participants will be randomly assigned to receive matched placebo (Days 0-13).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Suvorexant — Suvorexant is described chemically as: [(7R)-4-(5-chloro-2-benzoxazolyl) hexahydro-7-methyl-1H-1,4-diazepin-1-yl][5-methyl-2-(2H-1,2,3-triazol2-yl)phenyl]methanone. SUV's empirical formula is C23H23ClN6O2 and the molecular weight is 450.92. Each film coated tablet contains 10mg or 20mg of suvorexant.
  Other Names: SUV; Dual orexin receptor antagonist
  Arms: 10mg and 20mg Suvorexant (SUV)
Other: Placebo — Film coated tablet to match the active drug.
  Arms: Placebo

SUMMARY:
This study is to determine if suvorexant (SUV) will reduce insomnia in 76 men and women veteran and non-veterans between the ages 21-65 with posttraumatic stress disorder (PTSD) symptoms and alcohol use disorder (AUD). All participants will have a 7-day placebo run-in period, followed by a random assignment to receive placebo or suvorexant for an additonal 14 days. Post-randomization, participants will attempt to stop drinking for two weeks and will complete daily virtual diaries and study outcome assessments via in-person clinic visits on days 7 and 14.

DETAILED DESCRIPTION:
This is a randomized, double-masked, placebo-controlled study to evaluate preliminary efficacy and safety of suvorexant (SUV) (20mg) for sleep disturbance in alcohol use disorder (AUD) and co-occurring posttraumatic stress disorder (PTSD) symptoms in approximately 76 randomized men and women veteran and non-veterans between the ages 21-65. Participants will be recruited from the University of Texas Health Science Center at Houston (UTHealth) Trauma and Recovery Center (TRC) and the University of California - Los Angeles (UCLA) (in collaboration with West Los Angeles VA Medical Center). Following a 7-day placebo run-in, participants will be randomly assigned to receive SUV (10mg (Days 0-6) and 20mg (Days 7-13)) or matched placebo. Randomization will be stratified on sex and level of sleep disturbance (Insomnia Severity Index (ISI) score). Post-randomization, all participants will complete an alcohol cue-reactivity paradigm prior to the initial dose of study medication. The alcohol cue-reactivity paradigm is an established laboratory assessment of craving during which participants are exposed to real alcohol and water cues in a bar laboratory setting. Participants will then take their first dose of medication. Participants will begin the real-world quit attempt, during which they will attempt to stop drinking for two weeks. Participants will complete daily virtual diaries and visits to assess sleep, past-day drinking, and alcohol craving. Participants will return to one of the clinical sites on study Day 14 to complete an alcohol cue-reactivity session to assess post-medication craving. PTSD symptoms will be assessed via Clinician-Administered PTSD Scale for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (CAPS-5) and Post-traumatic Stress Disorder Checklist for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (PCL-5) at baseline, at Day 7 and at Day 14 of treatment with SUV or matched placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21 and 65.
* Meet current (i.e., past 12-month at Day -7/-6) DSM-5 diagnostic criteria for moderate or severe AUD as determined by the MINI.
* Currently experiencing PTSD symptoms at screening (Day -7/-6) as indicated by PCL-5 cut-score > 30.
* Intrinsic motivation to reduce or quit drinking (defined as self-reported intention at screening to reduce or quit drinking within the next 6 months) and to receive PTSD treatment.
* Must have an ISI score equal to or > 7 (subthreshold insomnia). ISI score below 7 at screening will not be included or proceed beyond the screening day.
* Agree to abstain from all other sleep medications (starting at Day -7).
* Have a place to live in the 2 weeks prior to randomization (Day 0) and not be at risk that s/he will lose his/her housing in the next month.

Exclusion Criteria:

* A current (past 12-month at Day -7/-6) DSM-5 diagnosis via the MINI of substance use disorder for any substances other than alcohol, nicotine, or marijuana (< moderate level on DSM 5).
* A lifetime DSM-5 diagnosis via the MINI of schizophrenia, bipolar disorder, or psychotic disorder.
* Positive urine test for any recreational drugs other than marijuana at screening (Day -7/-6).
* Current clinically significant alcohol withdrawal (i.e., score ≥ 10 on the CIWA-Ar).
* Currently pregnant, nursing, or no reliable method of birth control (females only).
* Any clinically significant medical condition that would preclude safe participation in the study (e.g. narcolepsy, seizure disorder, or other clinically significant cardiovascular, hematologic, hepatic, renal, neurological, or endocrine disorders).
* Use of suvorexant (within 30 days of Day -7).
* Currently on prescription medication that contraindicates use of suvorexant (including moderate or strong Cytochrome P450 3A modulators (CYP3A inhibitors and inducers))
* Hepatic insufficiency (AST/ALT > 5x upper limit of normal (ULN)).
* Suicidal Ideation determined by greater than moderate Columbia Suicide Severity Rating Scale.
* Inability to provide evidence of 48-hour alcohol abstinence (self-report, BrAC, EtG) at Day 0 AND failure after second attempt at 48-hour abstinence.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index (ISI) score from baseline to Day 14. | Baseline (Day 0) and Day 14
  The Insomnia Severity Index (ISI) is a brief questionnaire to screen for insomnia in participants. A scoring system is used to identify what degree insomnia (if any detected) is affecting daily life and sleep patterns. A total score is derived by summing all seven items with a total score ranging from 0 to 28 (with higher scores indicative of worse insomnia symptoms).

SECONDARY OUTCOMES:
Change in cue-induced alcohol craving, as assessed by the Alcohol Urge Questionnaire (AUQ) during the alcohol condition, from baseline to day 14. | Baseline (Day 0) and Day 14
  The Alcohol Urge Questionnaire (AUQ) consists of eight statements about the respondent's feelings and thoughts about drinking as they are completing the questionnaire (i.e., right now). The respondent is asked to respond to each statement about alcohol craving via a 7-item Likert scale ranging from "strongly disagree" to "strongly agree." Each item is scored on a 1 to 7 scale (Strongly Disagree = 1 and Strongly Agree = 7). Items 2 and 7 are reverse scored. A total score is computed by averaging the item scores. Higher scores reflect greater craving.
Change in mean number of drinks per drinking day from baseline to Day 14. | Baseline (Day 0) and Day 14
  Timeline Follow Back (TLFB) is a calendar-based method of assessing drinking patterns used to document the frequency and amount of daily alcohol consumption per day. Participants are given a blank calendar covering the time interval to be re-constructed and are asked to reconstruct retrospectively their drinking behavior over that interval. The TLFB will be used to calculate the number of drinks per day and drinks per drinking day over the course of the study period.
Percent total days abstinent during the 14-day quit attempt period. | Baseline (Day 0) through Day 14
  Timeline Follow Back (TLFB) is a calendar-based method of assessing drinking patterns used to document the frequency and amount of daily alcohol consumption per day. Participants are given a blank calendar covering the time interval to be re-constructed and are asked to reconstruct retrospectively their drinking behavior over that interval. The TLFB will be used to document the total number of abstinent days over the course of the study period.
Change in the mean number of days abstinent during the medication period (day 0 through 14) compared to the 30-days prior (screening period). | Screening (30-days prior to baseline) and Baseline through Day 14
  Timeline Follow Back (TLFB) is a calendar-based method of assessing drinking patterns used to document the frequency and amount of daily alcohol consumption per day. Participants are given a blank calendar covering the time interval to be re-constructed and are asked to reconstruct retrospectively their drinking behavior over that interval. The TLFB will be used to document the number of days with and without drinking from 30-days prior to baseline and 14-days post randomization.
Change in PTSD total symptom severity score as measured by the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) from baseline to Day 14. | Baseline (Day 0) through Day 14
  Gold-standard in PTSD assessment. The CAPS-5 is a 30-item structured interview that can be used to make current (past month) diagnosis of PTSD, make lifetime diagnosis of PTSD, and assess PTSD symptoms over the past week. The symptom severity score ranges from 0 to 80 with higher score indicating worse PTSD symptoms.
Change in PTSD score as measured by the PTSD Checklist for DSM-5 (PCL-5) from baseline to Day 14. | Baseline (Day 0) through Day 14
  The PCL-5 is a 20-item self-report measure that assesses DSM-5-based criteria for PTSD symptoms. Each item is rated on a 5-point Likert-type scale (0 = Not at all; 4 = Extremely) that indicates how much the participant has been bothered by an identified "worst" stressful event in the past month. The PTSD score ranges from 0 to 80 with higher score indication worse PTSD symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Lane, PhD, Principal Investigator — The University of Texas Health Science Center, Houston; Lara Ray, PhD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - University of California - Los Angeles, Los Angeles, California
  - The University of Texas Health Science Center - Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ray LA, Nieto SJ, Miotto K, Mooney L, LeBeau R, Yoon JH, Schmitz JM, Acierno R, Bailey NW, Jenkins J, Vincent J, Nolen T, Hirsch S, Williams A, Lane SD. Suvorexant for alcohol use disorder and post-traumatic stress disorder: study protocol for a phase II randomized clinical trial. Trials. 2026 Feb 3. doi: 10.1186/s13063-026-09489-7. Online ahead of print. PMID 41630040